CLINICAL TRIAL: NCT03362281
Title: Efficacy and Safety of Intravenous IIaprazole for Peptic Ulcer Bleeding: A Randomized, Double-Blind, Omeprazole-Controlled, Multicenter, and Phase 3 Trail in China
Brief Title: Ilaprazole for the Treatment and Prevention of Peptic Ulcer Bleeding in Chinese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Livzon-IYI-Ⅲ
Record Dates: First submitted 2017-11-28; First posted 2017-12-05 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Peptic Ulcer Hemorrhage
Keywords: Peptic ulcer hemorrhage; Proton Pump Inhibitor
MeSH Terms: conditions — Peptic Ulcer Hemorrhage | interventions — ilaprazole; Omeprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ilaprazole (Experimental)
  Interventions: Drug: Ilaprazole; Drug: Ilaprazole tablet; Drug: amoxicillin and clarithromycin
- omeprazole (Active Comparator)
  Interventions: Drug: Omeprazole; Drug: Ilaprazole tablet; Drug: amoxicillin and clarithromycin

INTERVENTIONS:
Drug: Ilaprazole — 10 mg ilaprazole daily (at day 1-3) through intravenous infusion within 30min with first dose doubling.
  Arms: Ilaprazole
Drug: Omeprazole — 40 mg omeprazole twice daily (at day 1-3) through intravenous infusion within 30min.
  Arms: omeprazole
Drug: Ilaprazole tablet — Since 4th day, those patients were changed to take oral ilaprazole tablets 10mg each day till 30th day
Drug: amoxicillin and clarithromycin — The Patients who with helicobacter pylori infection were provided amoxicillin and clarithromycin as complimentary therapy for two weeks

SUMMARY:
The purpose of this phase study is to confirm the efficacy and safety by compare ilaprazole and omeprazole in the treatment and prevention of peptic ulcer bleeding. Patients with endoscopically diagnosed peptic ulcer bleeding were enrolled in a multi-center, stratified randomized, non-inferiority test, double-blind, parallel and positive-controlled trial. They were randomly assigned into two groups, ilaprazole and omeprazole, to be treated for up to 30 days. The primary endpoint was the hemostasis rate at the end of 72 hours. Secondary end points include ulcer staging changes within 72 hours, effective rate of hemostasis, hemostasis duration, average blood transfusion and rebleeding rate, etc.

DETAILED DESCRIPTION:
Patients with endoscopically diagnosed gastric and duodenal ulcer bleeding were randomly assigned into two groups, ilaprazole and omeprazole. 360 patients were administrated 10 mg ilaprazole daily (at day 1-3) through intravenous infusion within 30min with first dose doubling. Other 180 patients were administrated 40 mg omeprazole twice daily (at day 1-3) through intravenous infusion for 30min. Since 4th day, both group taken oral ilaprazole tablets 10mg each day till 30th day; And the Patients who with helicobacter pylori infection were provided amoxicillin and clarithromycin as complimentary therapy for two weeks. The efficacy of ilaprazole and omeprazole was evaluated by the primary endpointthe-hemostasis rate at the end of 72 hours in the total population, high-risk groups and low-risk groups and secondary end points including ulcer staging changes within 72 hours, effective rate of hemostasis, hemostasis duration, average blood transfusion, the need to switch to other treatments (endoscopic treatment or surgery, etc.), the disappearance time of ulcer pain and rebleeding rate. This phase Ⅲ clinical trial was designed to confirm the efficacy and safety of ilaprazole in the treatment of peptic ulcer bleeding and to pride a basis for registration.

ELIGIBILITY:
Inclusion Criteria:

1. were 18-70 years of age, male or female.
2. had symptoms of hematemesis, hematochezia, melena within 24 hours and clinically diagnosed as peptic ulcer bleeding.
3. had endoscopically diagnosed gastric or duodenal ulcer bleeding and 3mm ≤ ulcer diameter ≤ 15mm.
4. underwent local hemostasis according to "Acute non-variceal upper gastrointestinal bleeding guidelines (2009, Hangzhou)" Forrest grading; multiple ulcers was judged by the higher level.
5. voluntarily sign informed consent

Exclusion Criteria:

1. had hemorrhagic shock ( systolic blood pressure<90mmHg) or require surgery.
2. were non-ulcer bleeding and gastric ulcer biopsy proved malignant.
3. had gastrectomy and gastrointestinal anastomosis.
4. were suffering from serious heart, liver, brain, lung, kidney and other serious diseases.
5. had coagulation disorders (laboratory tests showed that platelets <80 × 109 / L, PT abnormal and exceed the normal control for 3 seconds, APTT than the normal control for 10 seconds).
6. had hypersensitivity or idiosyncratic reaction to ilaprazole, omeprazole, esomeprazole or any other benzimidazole.
7. had positive result of urine pregnancy test.
8. used the same kind of drugs within 48 hours before entering the group.
9. need to continue the combination of the following drugs that have an effect on treatment during the study: NSAIDs, corticosteroids, heparin, warfarin and vitamin K, platelet antagonists or other hemostatic agents.
10. participated in a clinical trial with an investigational drug or device within the past three months.
11. had alcoholic intemperance, drug addiction or other factors that researchers think it unfit for drug clinical trials.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
the rate of hemostasis | 72 hours
  the hemostasis rate checked by endoscopy within 72 hours